CLINICAL TRIAL: NCT07325799
Title: Evaluation of the Association Between Anesthesia Type and Postoperative Sleep Quality in Septoplasty Patients: A Prospective Observational Study
Brief Title: Anesthesia Type and Postoperative Sleep Quality in Septoplasty
Acronym: ANES-SLEEP
Status: Recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Sevim Şenol Karataş, Anesthesiology and Reanimation Specialist, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSH-ANES-SEP-SLEEP-2025
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Sleep Quality; Nasal Septum Deviation; Septoplasty; Total Intravenous Anesthesia; Inhalational Anesthesia
Keywords: Total Intravenous Anesthesia; Inhalational Anesthesia; Postoperative Sleep Quality; Richards-Campbell Sleep Questionnaire; Septoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Intravenous Anesthesia: Patients receiving total intravenous anesthesia as part of routine clinical practice.
- Inhalational Anesthesia: Patients receiving inhalational general anesthesia according to routine clinical practice.

SUMMARY:
This prospective observational study aims to evaluate the association between routinely applied anesthesia techniques and postoperative sleep quality in adult patients undergoing septoplasty. Patients will receive either total intravenous anesthesia or inhalational anesthesia according to standard clinical practice, without any intervention by the investigators. Postoperative sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire on postoperative days 7 and 15. Secondary outcomes include postoperative pain intensity, opioid consumption, and postoperative nausea and vomiting.

DETAILED DESCRIPTION:
This study is designed as a prospective, observational cohort study conducted at a single tertiary care center. The study population will consist of adult patients undergoing elective septoplasty for nasal septum deviation. All patients will receive general anesthesia as part of routine clinical care, either using total intravenous anesthesia (TIVA) or inhalational anesthesia, according to the anesthesiologist's standard practice. No randomization or study-related intervention will be performed.

Eligible patients will be enrolled consecutively after providing written informed consent. Demographic data, clinical characteristics, American Society of Anesthesiologists (ASA) physical status, duration of surgery, anesthesia technique, perioperative opioid consumption, and postoperative complications will be recorded prospectively using hospital electronic medical records and standardized case report forms.

Postoperative sleep quality will be evaluated using the Richards-Campbell Sleep Questionnaire (RCSQ), a validated patient-reported outcome measure. Follow-up assessments will be conducted via telephone interviews on postoperative days 7 and 15. Pain intensity will be assessed using the Numerical Pain Rating Scale, and postoperative nausea and vomiting will be evaluated using a standardized ordinal scale.

ELIGIBILITY:
Inclusion Criteria:

* - Adults aged 18 years and older
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective septoplasty under general anesthesia
* Willing and able to provide written informed consent
* Agree to postoperative follow-up telephone interviews on postoperative days 7 and 15

Exclusion Criteria:

* - ASA physical status IV or V
* Age younger than 18 years
* Severe obstructive sleep apnea confirmed by polysomnography and requiring active CPAP therapy
* Significant cognitive impairment, delirium, or active psychiatric disorder preventing reliable questionnaire completion
* Chronic use of opioids, benzodiazepines, hypnotics, sedatives, or antipsychotic medications (≥3 days per week within the last month)
* Alcohol or substance abuse
* Major intraoperative complications, unplanned intensive care unit admission, or reoperation within the first 24 hours
* Pregnancy or breastfeeding
* Severe systemic disease or unstable cardiopulmonary condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years and older who are scheduled to undergo elective septoplasty under general anesthesia. Patients will receive either total intravenous anesthesia or inhalational anesthesia according to routine clinical practice. Only patients who provide written informed consent and agree to postoperative follow-up assessments will be included. The study population will be recruited from a single tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire (RCSQ) Total Score | Postoperative day 7 and postoperative day 15
  Postoperative sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ).
  The total RCSQ score ranges from 0 to 100 and is calculated as the mean of five core items.
  Higher scores indicate better sleep quality.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | Postoperative day 7 and postoperative day 15
  Postoperative pain intensity will be assessed using the Numerical Pain Rating Scale, ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Lin D, Huang X, Sun Y, Wei C, Wu A. Perioperative Sleep Disorder: A Review. Front Med (Lausanne). 2021 Jun 7;8:640416. doi: 10.3389/fmed.2021.640416. eCollection 2021. PMID 34164409
- [Background] Li S, Song B, Li Y, Zhu J. Effects of Intravenous Anesthetics vs Inhaled Anesthetics on Early Postoperative Sleep Quality and Complications of Patients After Laparoscopic Surgery Under General Anesthesia. Nat Sci Sleep. 2021 Mar 15;13:375-382. doi: 10.2147/NSS.S300803. eCollection 2021. PMID 33758567